CLINICAL TRIAL: NCT03203525
Title: A Phase I Study of the NovoTTF-100L(P) System to Enhance Antitumor Activity in Patients With Predominant Hepatic Metastatic Cancer
Brief Title: Combination Chemotherapy and Bevacizumab With the NovoTTF-100L(P) System in Treating Participants With Advanced, Recurrent, or Refractory Hepatic Metastatic Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-0357; NCI-2018-01597 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2014-0357 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2017-06-27; First posted 2017-06-29 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Advanced Malignant Neoplasm; Colorectal Carcinoma Metastatic in the Liver; Metastatic Malignant Neoplasm in the Liver; Refractory Malignant Neoplasm
MeSH Terms: conditions — Neoplasms | interventions — Bevacizumab; Immunoglobulin G; Disulfides; Fluorouracil; dehydroftorafur; Leucovorin; Oxaliplatin; liposomal doxorubicin; Doxorubicin; temsirolimus; Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (FOLFOX6, bevacizumab, NovoTTF-100L[P]) (Experimental): Participants receive oxaliplatin, leucovorin, and fluorouracil via pump over 46 hours on beginning on day 1, bevacizumab IV over 30-90 minutes on days 1 and 15, and use NovoTTF-100L(P) system over 18 hours daily. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Bevacizumab; Drug: Fluorouracil; Drug: Leucovorin; Drug: Oxaliplatin; Procedure: Tumor Treating Fields Therapy
- Arm B(bevacizumab,liposomal doxorubicin, DAT, NovoTTF-100L[P]) (Experimental): Participants receive bevacizumab IV over 90 minutes on days 1 and 15, pegylated liposomal doxorubicin hydrochloride IV over 30 minutes-3 hours on days 1 and 15, and temsirolimus IV over 60-90 minutes on days 1, 8, 15, and 22. Participants also use NovoTTF-100L(P) system over 18 hours daily. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Bevacizumab; Drug: Pegylated Liposomal Doxorubicin Hydrochloride; Drug: Temsirolimus; Procedure: Tumor Treating Fields Therapy

INTERVENTIONS:
Biological: Bevacizumab — Given IV
  Other Names: Anti-VEGF; Anti-VEGF Humanized Monoclonal Antibody; Anti-VEGF rhuMAb; Avastin; Bevacizumab awwb; Bevacizumab Biosimilar BEVZ92; Bevacizumab Biosimilar BI 695502; Bevacizumab Biosimilar CBT 124; Bevacizumab Biosimilar CT-P16; Bevacizumab Biosimilar FKB238; Bevacizumab Biosimilar HD204; Bevacizumab Biosimilar HLX04; Bevacizumab Biosimilar IBI305; Bevacizumab Biosimilar LY01008; Bevacizumab Biosimilar MIL60; Bevacizumab Biosimilar QL 1101; Bevacizumab Biosimilar RPH-001; Bevacizumab Biosimilar SCT501; BP102; BP102 Biosimilar; HD204; Immunoglobulin G1 (Human-Mouse Monoclonal rhuMab-VEGF Gamma-Chain Anti-Human Vascular Endothelial Growth Factor), Disulfide With Human-Mouse Monoclonal rhuMab-VEGF Light Chain, Dimer; Recombinant Humanized Anti-VEGF Monoclonal Antibody; rhuMab-VEGF; SCT501
Drug: Fluorouracil — Given via pump
  Other Names: 5 Fluorouracil; 5 Fluorouracilum; 5 FU; 5-Fluoro-2,4(1H, 3H)-pyrimidinedione; 5-fluorouracil; 5-Fluracil; 5-FU; 5FU; AccuSite; Carac; Fluoro Uracil; Fluouracil; Flurablastin; Fluracedyl; Fluracil; Fluril; Fluroblastin; Ribofluor; Ro 2-9757; Ro-2-9757
  Arms: Arm A (FOLFOX6, bevacizumab, NovoTTF-100L[P])
Drug: Leucovorin — Given via pump
  Other Names: folinic acid
  Arms: Arm A (FOLFOX6, bevacizumab, NovoTTF-100L[P])
Drug: Oxaliplatin — Given via pump
  Other Names: 1-OHP; Ai Heng; Aiheng; Dacotin; Dacplat; Diaminocyclohexane Oxalatoplatinum; Eloxatin; Eloxatine; JM-83; Oxalatoplatin; Oxalatoplatinum; RP 54780; RP-54780; SR-96669
  Arms: Arm A (FOLFOX6, bevacizumab, NovoTTF-100L[P])
Drug: Pegylated Liposomal Doxorubicin Hydrochloride — Given IV
  Other Names: ATI-0918; Caelyx; DOX-SL; Doxil; Doxilen; Doxorubicin HCl Liposomal; Doxorubicin HCl Liposome; Doxorubicin Hydrochloride Liposome; Duomeisu; Evacet; LipoDox; Lipodox 50; Liposomal Adriamycin; Liposomal Doxorubicin Hydrochloride; Liposomal-Encapsulated Doxorubicin; Pegylated Doxorubicin HCl Liposome; S-Liposomal Doxorubicin; Stealth Liposomal Doxorubicin; TLC D-99
  Arms: Arm B(bevacizumab,liposomal doxorubicin, DAT, NovoTTF-100L[P])
Drug: Temsirolimus — Given IV
  Other Names: CCI-779; CCI-779 Rapamycin Analog; Cell Cycle Inhibitor 779; Rapamycin Analog; Rapamycin Analog CCI-779; Torisel
  Arms: Arm B(bevacizumab,liposomal doxorubicin, DAT, NovoTTF-100L[P])
Procedure: Tumor Treating Fields Therapy — Use NovoTTF-100L(P) system
  Other Names: Alternating Electric Field Therapy; TTF; TTFields

SUMMARY:
This phase I trial studies the side effects and best dose of combination chemotherapy and bevacizumab, and to see how well they work with the NovoTTF-100L(P) system in treating participants with cancer that has come back or does not respond to treatment and has spread to the liver. Drugs used in chemotherapy, such as oxaliplatin, leucovorin, fluorouracil, pegylated liposomal doxorubicin hydrochloride, and temsirolimus, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Bevacizumab is a monoclonal antibody that may interfere with the ability of tumor cells to grow and spread. The NovoTTF-100L(P) system is a portable device that uses electrical fields to stop the growth of tumor cells. Giving combination chemotherapy and monoclonal antibody therapy while using the NovoTTF-100L(P) system may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To define the maximum tolerated doses (MTD) of two established chemotherapy regimens (Arm A: FOLFOX6 [oxaliplatin, fluorouracil (5FU) and leucovorin (folinic acid)] plus bevacizumab; and Arm B: pegylated liposomal doxorubicin hydrochloride [liposomal doxorubicin] and bevacizumab plus temsirolimus [DAT]) in combination with the concurrent use of the NovoTTF-100L(P) system in patients with predominant hepatic metastases.

II. To define the safety profiles of FOLFOX6 plus bevacizumab or DAT with concurrent NovoTTF-100L(P) in patients with predominant hepatic metastases.

SECONDARY OBJECTIVES:

I. To evaluate clinical response signals to the treatment with FOLFOX6 plus bevacizumab or DAT with concurrent NovoTTF-100L(P).

II. To assess predictive biomarkers by analyzing baseline molecular mutation status, and resistant pathways by comparing molecular signatures at baseline versus at time of relapse in patients who have achieved objective responses.

OUTLINE: This is a dose-escalation study. Participants are assigned to 1 of 2 arms.

ARM A: Participants receive oxaliplatin, leucovorin, and fluorouracil via pump over 46 hours beginning on day 1, bevacizumab intravenously (IV) over 30-90 minutes on days 1 and 15, and use NovoTTF-100L(P) system over 18 hours daily. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ARM B: Participants receive bevacizumab IV over 90 minutes on days 1 and 15, pegylated liposomal doxorubicin hydrochloride IV over 30 minutes-3 hours on days 1 and 15, and temsirolimus IV over 60-90 minutes on days 1, 8, 15, and 22. Participants also use NovoTTF-100L(P) system over 18 hours daily. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After the completion of study treatment, patients are followed at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced malignancies, either refractory to standard therapy or for which no effective standard therapy is available, unless the drugs in the protocol are part of the standard of care for a specific diagnosis

  * Predominant hepatic metastasis is defined as at least 50% of the total tumor burden involving the liver
  * An aberrant PI3K pathway such as PIK3CA mutations or PTEN loss, is detected in a CLIA (Clinical Laboratory Improvement Amendments)-certified laboratory
  * For patients who are enrolled into the arm of FOLFOX6 plus bevacizumab, they must have metastatic colorectal cancer with predominant hepatic metastases
  * For patients who are enrolled into the arm of DAT, they must have predominant hepatic metastases harboring an aberrant PI3K pathway
* Patients must have measurable or evaluable disease, as defined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
* Women of child-bearing potential (women who are not postmenopausal for at least one year or are not surgically sterile) and men must agree to use adequate contraception (e.g., hormonal, barrier device, or abstinence) prior to study entry, for the duration of study participation, and for 30 days after the last dose of the study agents
* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2
* Neutrophils >= 1,500/uL
* Platelets >= 100,000/uL
* Total bilirubin =< 1.5 x ULN (upper limit of normal) (except patients with Gilbert's syndrome, who must have a total bilirubin =< 3.0 mg/dL)
* Alanine aminotransferase (ALT) =< 3 x ULN or =< 5 x ULN if liver metastases persist
* Serum creatinine =< 1.5 mg/dL or calculated creatinine clearance >= 50 mL/minutes
* Patients should be able to read and fully understand the requirements of the trial, be willing to comply with all trial visits and assessments, and be willing and able to sign an Institutional Reviewed Board (IRB)-approved written informed consent document
* Patients may receive palliative radiation therapy immediately before or during the treatment if the radiation therapy is not delivered to the sole target lesions

Exclusion Criteria:

* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection requiring intravenous antibiotics, symptomatic congestive heart failure (New York Heart Association [NYHA] class III or IV), unstable angina pectoris, uncontrolled systemic hypertension (systolic blood pressure [BP] > 140 mm Hg, diastolic BP > 90 mm Hg), left ventricular ejection fraction < 50%, active bleeding, or psychiatric illness/social situations that would limit compliance with study requirements
* Patients who have not recovered from major surgical procedure, or significant traumatic injury (i.e., patients still need additional medical care for these issues)
* History of allergic reactions to the study drugs or their analogs, or any component of the products, or sensitive to conductive hydrogels used on electrocardiogram (ECG) stickers or transcutaneous electrical nerve stimulation (TENS) electrodes
* Any treatment specific for tumor control within 3 weeks of drugs; or within 2 weeks if cytotoxic agents were given weekly (within 6 weeks for nitrosoureas or mitomycin C), or within 5 half-lives for targeted agents with half-lives and pharmacodynamic effects lasting fewer than 4 days (that includes, but is not limited to, erlotinib, sorafenib, sunitinib, bortezomib, and similar agents), or failure to recover from the toxic effect of any of these therapies prior to study entry
* Symptomatic primary tumors or metastasis of brain and/or central nervous system that are uncontrolled with antiepileptics and requiring high doses of steroids
* Implanted pacemaker, defibrillator, nerve stimulator or other active electronic medical devices
* Corrected QT interval (QTc) is greater than 480 milliseconds (msec) at screening, or documented clinically significant arrhythmias. The QTc formula Bazett will be used for assessing subject eligibility
* History of stroke or transient ischemic attack, peripheral vascular disease, active gastric or duodenal ulcer, abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to study enrollment
* Patients with known human immunodeficiency virus infection, active hepatitis B or C
* Women who are pregnant will be excluded from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2020-06-23 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 3 years
  Descriptive statistics will be provided on the grade and type of toxicity by dose level.

SECONDARY OUTCOMES:
Response | Up to 3 years
  Will be assessed by Response Evaluation Criteria in Solid Tumors 1.1. Wilcoxon's Signed-Rank Test and Fisher's exact test will be used for data analysis of continuous variables and categorical variables, respectively. A mixed model accounting for patient effects will be used to analyze longitudinal data (including biomarker data) over time.
Biomarker analysis | Up to 3 years
  Wilcoxon's Signed-Rank Test and Fisher's exact test will be used for data analysis of continuous variables and categorical variables, respectively. A mixed model accounting for patient effects will be used to analyze longitudinal data (including biomarker data) over time.

CONTACTS AND LOCATIONS:
Overall Officials: Siqing Fu, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org